CLINICAL TRIAL: NCT00193219
Title: A Randomized Phase II Study of Modified FOLFOX6 (Infusional 5-Fluorouracil/Leucovorin, Oxaliplatin) and Bevacizumab With or Without Cetuximab in Patients With Metastatic Colorectal Cancer
Brief Title: Bevacizumab and Cetuximab in Combination With FOLFOX6 in Patients With Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI GI 64
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Results first posted 2013-03-07 (Estimated); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Colon Cancer
Keywords: Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms | interventions — Bevacizumab; Cetuximab; Fluorouracil; Leucovorin; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Experimental): Bevacizumab 5 mg/kg IV
  Cetuximab 400 mg/m2 (first cycle only) IV on day 1 and 250 mg/m2 IV on day 8 with all subsequent cycles 250 mg/m2 IV on days 1 and 8
  5-Fluorouracil 400 mg/m2 bolus IV bolus followed by 2400 mg/m2 administered as continuous IV infusion over 46 hours via pump (outpatient)
  Leucovorin 350 mg IV
  Oxaliplatin 85 mg/m2 IV
  Interventions: Drug: Bevacizumab; Drug: Cetuximab; Drug: 5-fluorouracil; Drug: Leucovorin; Drug: Oxaliplatin

INTERVENTIONS:
Drug: Bevacizumab — 5 mg/kg IV
  Other Names: Avastin
Drug: Cetuximab — 400 mg/m2 (first cycle only) IV on day 1 and 250 mg/m2 IV on day 8 with all subsequent cycles 250 mg/m2 IV on days 1 and 8
  Other Names: Erbitux
Drug: 5-fluorouracil — 400 mg/m2 bolus IV bolus followed by 2400 mg/m2 administered as continuous IV infusion over 46 hours via pump (outpatient)
  Other Names: 5-FU; Adrucil
Drug: Leucovorin — 350 mg IV
  Other Names: Folinic Acid
Drug: Oxaliplatin — 85 mg/m2 IV
  Other Names: Eloxatin

SUMMARY:
This trial will evaluate the combination of modified infusional 5-fluorouracil/ leucovorin, oxaliplatin (FOLFOX6), bevacizumab, and cetuximab in patients with metastatic colorectal cancer. FOLFOX6 has proven to be a safe and effective regimen in first line treatment of advanced colorectal cancer. The role of epidermal growth factor (EGFR) inhibitors in an earlier treatment setting in combination with optimal chemotherapy regimens is an important emerging question.

DETAILED DESCRIPTION:
All patients received cetuximab: 400 mg/m2 (first cycle only) administered intravenously (IV) on day 1 and 250 mg/m2 IV on day 8 with all subsequent cycles 250 mg/m2 IV on days 1 and 8. Day 1 cetuximab was immediately followed by bevacizumab 5 mg/kg IV, oxaliplatin 85 mg/m2 IV, and 5-fluorouracil 400 mg/m2 IV bolus, followed by 2400 mg/m2 administered as a continuous infusion over 46 hours via a pump (outpatient) and leucovorin 350 mg IV (modified FOLFOX6). Cycles were 14 days.

ELIGIBILITY:
Inclusion Criteria:

To be included in the study, you must meet the following criteria:

* Metastatic colorectal cancer confirmed by a biopsy sample
* 18 years of age or older
* Evidence of disease progression at time of study entry
* At least one prior adjuvant chemotherapy regimen
* No prior therapy for metastatic disease
* Measurable disease
* Able to perform activities of daily living with minimal assistance
* Adequate bone marrow, kidney, and liver function
* Tumor tissue available for assessment of EGFR
* Signed informed consent

Exclusion Criteria:

You cannot participate in the study if any of the following apply to you:

* Treatment with a previous regimen for metastatic disease
* Prior treatment with any EGFR inhibitor or anti-angiogenic agents
* Brain or nervous system metastases
* History of severe thromboembolic event
* Clinical evidence or history of bleeding or coagulopathy
* History of stroke or heart attack within six months
* Poorly controlled hypertension
* Non-healing wound, ulcer, or bone fracture
* History of abdominal fistula, perforation, or abscess within six months
* Other uncontrolled or significant disease or medical condition

Please note: There are additional inclusion/exclusion criteria. The study center will determine if you meet all of the criteria. If you do not qualify for the trial, study personnel will explain the reasons. If you do qualify, study personnel will explain the trial in detail and answer any questions you may have. You can then decide if you wish to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2005-07; Primary Completion 2008-06 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David R. Spigel, MD, Principal Investigator — SCRI Development Innovations, LLC
Locations (10):
- United States (10):
  - Oncology Hematology Associates of SW Indiana, Evansville, Indiana
  - Consultants in Blood Disorders and Cancer, Louisville, Kentucky
  - Mercy Hospital, Portland, Maine
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - Jackson Oncology Associates, Jackson, Mississippi
  - St. Louis Cancer Care, Chesterfield, Missouri
  - Methodist Cancer Center, Omaha, Nebraska
  - Oncology Hematology Care, Cincinnati, Ohio
  - Chattanooga Oncology and Hematology Associates, Chattanooga, Tennessee
  - Tennessee Oncology, Nashville, Tennessee

REFERENCES:
- [Background] Spigel DR, Greco FA, Waterhouse D, Shipley D, Lane CM, Vazquez ER, Clark BL, Infante JR, Bendell JC, Burris HA 3rd, Hainsworth JD. Phase II trial of FOLFOX6, bevacizumab, and cetuximab in the first-line treatment of metastatic colorectal cancer. Clin Adv Hematol Oncol. 2010 Jul;8(7):480-5, 498. PMID 20864916
- See also: Related Info — http://www.clinicaladvances.com/index.php/our_publications/hem_onc-article/1739/

RESULTS

PARTICIPANT FLOW:
Groups:
- Bevacizumab/Cetuximab/FOLFOX: Bevacizumab 5 mg/kg IV Cetuximab 400 mg/m2 (first cycle only) IV on day 1 and 250 mg/m2 IV on day 8 with all subsequent cycles 250 mg/m2 IV on days 1 and 8 5-Fluorouracil 400 mg/m2 bolus IV bolus followed by 2400 mg/m2 administered as continuous IV infusion over 46 hours via pump (outpatient) Leucovorin 350 mg IV Oxaliplatin 85 mg/m2 IV
Period: Overall Study
Arm/Group | Bevacizumab/Cetuximab/FOLFOX
Started | 36
Completed | 6
Not Completed | 30

BASELINE CHARACTERISTICS:
Arm/Group | Bevacizumab/Cetuximab/FOLFOX
Number analyzed (Participants) | 36
Age, Continuous [Median (Full Range); unit: years] | 55 [29 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 20
Region of Enrollment [Number; unit: participants]
  United States | 36

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR), the Percentage of Patients Who Experience an Objective Benefit From Treatment
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI or CT: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 18 months
Population: This study was originally designed as a randomized study with patients receiving FOLFOX and bevacizumab with or without cetuximab. Following an amendment, all patients received cetuximab, FOLFOX and bevacizumab. The 5 patients randomized prior to the amendment that did not receive cetuximab are excluded from the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Bevacizumab/Cetuximab/FOLFOX
Number analyzed (Participants) | 31
percentage of patients | 55 [36 to 73]

2. Secondary Outcome: Progression Free Survival (PFS), the Length of Time, in Months, That Patients Were Alive From Their First Date of Protocol Treatment Until Worsening of Their Disease
Description: Progression Free Survival (PFS) is defined as the interval between the start date of treatment and the date of occurrence of progressive disease or death.
Time Frame: 18 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab/Cetuximab/FOLFOX
Number analyzed (Participants) | 31
months | 9 [8.3 to 15.2]

3. Secondary Outcome: Overall Survival (OS), the Length of Time, in Months, That Patients Were Alive From Their First Date of Protocol Treatment Until Death
Description: Measured from the date of first treatment until the date of death from any cause
Time Frame: 36 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab/Cetuximab/FOLFOX
Number analyzed (Participants) | 31
months | 25.7 [15.4 to 27.6]

4. Secondary Outcome: Number of Patients With Adverse Events as a Measure of Safety With FOLFOX6 Combined With Bevacizumab and Cetuximab
Description: The toxicity assessments were made according to the common terminology criteria for adverse events (CTCAE version 3.0) of the National Cancer Institute. Number of participants with Grade 1 to 5 adverse events are reported here.
Time Frame: 18 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Bevacizumab/Cetuximab/FOLFOX
Number analyzed (Participants) | 31
Participants | 31

ADVERSE EVENTS:
Groups:
- Bevacizumab/FOLFOX: Bevacizumab 5 mg/kg IV; Fluorouracil 400 mg/m2 bolus IV bolus followed by 2400 mg/m2 administered as continuous IV infusion over 46 hours via pump (outpatient); Leucovorin 350 mg IV; Oxaliplatin 85 mg/m2 IV
Arm/Group | Bevacizumab/Cetuximab/FOLFOX | Bevacizumab/FOLFOX
Serious Adverse Events (participants affected / at risk) | 14/31 | 2/5
Other Adverse Events (participants affected / at risk) | 31/31 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bevacizumab/Cetuximab/FOLFOX (N=31) | Bevacizumab/FOLFOX (N=5)
Pain - Gastrointestinal (Gastrointestinal disorders) | 2 (2) | 0 (0)
Thrombosis/Thrombus/Embolism (Vascular disorders) | 4 (4) | 0 (0)
Hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dehydration (Gastrointestinal disorders) | 1 (1) | 0 (0)
ARDS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Mental Status (Nervous system disorders) | 1 (1) | 0 (0)
Pain - Abdominal (Gastrointestinal disorders) | 1 (1) | 0 (0)
Progressive Disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Pain - Renal/Genitourinary (Renal and urinary disorders) | 1 (1) | 0 (0)
Dementia (Psychiatric disorders) | 1 (1) | 0 (0)
Blurred Vision (Eye disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Venous Occlusion (Vascular disorders) | 1 (1) | 0 (0)
Allergic Reaction (Immune system disorders) | 2 (2) | 0 (0)
Febrile Neutropenia (Infections and infestations) | 1 (1) | 0 (0)
Multi Organ Failure (General disorders) | 1 (1) | 0 (0)
Chemoport Malfunction (Surgical and medical procedures) | 1 (1) | 0 (0)
Acute Appendicitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hearing loss (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bevacizumab/Cetuximab/FOLFOX (N=31) | Bevacizumab/FOLFOX (N=5)
Alopecia (Skin and subcutaneous tissue disorders) | 11 (54) | 1 (1)
Altered Mental Status (Nervous system disorders) | 2 (3) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 19 (105) | 3 (45)
Anorexia (Gastrointestinal disorders) | 22 (83) | 1 (4)
Anxiety (Psychiatric disorders) | 3 (6) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (13) | 1 (1)
Blurred Vision (Eye disorders) | 2 (4) | 0 (0)
Chills (General disorders) | 4 (8) | 0 (0)
Cold Sensitivity (General disorders) | 8 (36) | 2 (4)
Confusion (Nervous system disorders) | 2 (3) | 0 (0)
Constipation (Gastrointestinal disorders) | 14 (52) | 2 (7)
Cramps (abdominal) (Gastrointestinal disorders) | 2 (3) | 0 (0)
Deep Vein Thrombosis (Blood and lymphatic system disorders) | 3 (21) | 0 (0)
Dehydration (Gastrointestinal disorders) | 3 (4) | 0 (0)
Depression (Psychiatric disorders) | 4 (6) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 22 (112) | 3 (14)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (8) | 0 (0)
Dysuria (Renal and urinary disorders) | 3 (5) | 0 (0)
Edema (Blood and lymphatic system disorders) | 8 (21) | 0 (0)
Elevated AST (Hepatobiliary disorders) | 2 (3) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 2 (6)
Esophagitis (Infections and infestations) | 3 (5) | 0 (0)
Fatigue (General disorders) | 30 (248) | 5 (37)
Febrile Neutropenia (Infections and infestations) | 3 (7) | 0 (0)
Fever (General disorders) | 6 (9) | 1 (1)
Fingertip Fissures (Skin and subcutaneous tissue disorders) | 2 (12) | 0 (0)
Flu Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3)
Hemorrhoids (Gastrointestinal disorders) | 4 (15) | 0 (0)
Hiccoughs (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 11 (36) | 0 (0)
Hypersensitivity Reaction (General disorders) | 5 (5) | 1 (12)
Hypertension (Cardiac disorders) | 2 (4) | 1 (6)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (8) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 4 (6) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 3 (10) | 0 (0)
Indigestion (Gastrointestinal disorders) | 2 (2) | 0 (0)
Infection (Infections and infestations) | 3 (4) | 0 (0) — Infection not otherwise specified
Infection (Infections and infestations) | 2 (2) | 0 (0) — Sinus
Insomnia (General disorders) | 7 (13) | 2 (22)
leukopenia (Blood and lymphatic system disorders) | 19 (76) | 0 (0)
Motor Neuropathy (Nervous system disorders) | 0 (0) | 1 (8)
Mucositis (Gastrointestinal disorders) | 13 (35) | 2 (12)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Nail Changes (Skin and subcutaneous tissue disorders) | 4 (16) | 1 (1)
Nausea (Gastrointestinal disorders) | 24 (75) | 2 (18)
Neutropenia (Blood and lymphatic system disorders) | 25 (92) | 4 (34)
Night Sweats (General disorders) | 0 (0) | 1 (3)
Pain (General disorders) | 20 (80) | 3 (16)
palmar plantar erythrodysesthesia (Skin and subcutaneous tissue disorders) | 5 (16) | 0 (0)
Proteinuria (Metabolism and nutrition disorders) | 12 (30) | 1 (4)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 (12) | 0 (0)
reflux (Gastrointestinal disorders) | 2 (7) | 0 (0)
Sensory Neuropathy (Nervous system disorders) | 20 (136) | 3 (36)
Sinus Drainage (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
sinus infection (Infections and infestations) | 2 (2) | 0 (0)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 4 (17) | 0 (0)
Taste Alteration (Gastrointestinal disorders) | 7 (19) | 0 (0) — Dysgeusia
thrombocytopenia (Blood and lymphatic system disorders) | 19 (78) | 0 (0)
Vomiting (Gastrointestinal disorders) | 14 (28) | 2 (3)
Weakness (General disorders) | 7 (34) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review/embargo results communications prior to public release for a period that is >60 days but ≤180 days from date submitted to sponsor, who may require changes to the communication in order to remove specifically identified confidential information (other than study data) and/or delay the proposed publication to enable the sponsor to seek patent protection for inventions. The PI may not publish its results until 18 mos. after the trial has been completed at all sites.